CLINICAL TRIAL: NCT04390633
Title: Qualitative Assessment of the Needs and Knowledge of Patients With Chronic Intestinal Failure of Their Disease as Well as Those of Their Practitioners
Brief Title: Perception of Needs of Patients With Chronic Intestinal Failure and Their Practitioners: a Qualitative Study
Acronym: SBS-NEEDS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Société Francophone Nutrition Clinique et Métabolisme (Other)
Responsible Party: Sponsor
Other Study IDs: EI/2019/616
Record Dates: First submitted 2020-05-11; First posted 2020-05-15 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-03

CONDITIONS: Chronic Intestinal Failure; Small Intestine Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SBS NEEDS Study is a qualitative transversal study aiming to describe and understand the needs and knowledge of patients with Chronic Intestinal Failure as well as the representations of their practitioners

Chronic Intestinal Failure (CIF) is the long-lasting reduction of gut function, below the minimum necessary for the absorption of macronutrients and/or water and electrolytes, such that intravenous supplementation is required to maintain health and/or growth. CIF is the rarest organ failure. Home parenteral nutrition (HPN) is the primary treatment for CIF.

Semi-structured interviews will be conducted with patients in two nutrition unit and specialized in the small bowel diseases in two French region. 20 situations will be included.

After analysing the data of the individual interviews, focus groups will be conducted with health professionals from an accredited home parenteral nutrition department.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and over
* With Chronic Intestinal Failure (CIF) : "reduction of the intestinal functional mass below the minimum mass sufficient to ensure the absorption of nutrients to maintain nutritional status"
* medical follow-up in one of the two nutrition departments of the study
* Informed consent stating that the subject understood the purpose and methodology of the study and agrees to participate in the study.

Exclusion Criteria:

* Persons with proven and significant cognitive impairment preventing the completion of semi-structured interviews
* Person who does not speak French easily
* Generally, any person unlikely to cooperate in the study
* Adults under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women aged 18 and over, fulfilling the conditions of major Chronic Intestinal Failure (CIF) : "reduction of the intestinal functional mass below the minimum mass sufficient to ensure the absorption of nutrients to maintain nutritional status"
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
20 semi-structured interviews | 12 months
  Qualitative data analysis - Theorical saturation